CLINICAL TRIAL: NCT05096130
Title: The Effect of Lifestyle Modifications on Aspects Related to Fatigue, Quality of Life, Health, and Sleepiness in Professional Drivers
Brief Title: Lifestyle Medicine Strategies for Combating Sleepiness and Fatigue in Professional Drivers
Acronym: HighWay2Health
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Giorgos K. Sakkas, Ass Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1818/09/06/2021
Record Dates: First submitted 2021-09-30; First posted 2021-10-27 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Sleepiness, Daytime; Fatigue; Sleep Disorders, Circadian Rhythm
Keywords: driving; lifestyle medicine; Quality of life; Physical Activity; Diet; stress; sleep coaching; road accidents
MeSH Terms: conditions — Disorders of Excessive Somnolence; Fatigue; Sleep Disorders, Circadian Rhythm; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial. The study is composed of two groups. Group 1 is the control group and Group 2 is the experimental one. The trial period will last for 6 months for both groups. Intervention includes lifestyle changes targeting physical activity, diet, stress and sleep quality. The design is parallel.
Who Masked: Outcomes Assessor
Masking Description: Parameters such as questionnaires' scores, polysomnography outcomes, indices of health, and other data will be masked and coded for blind analysis by the main investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group - No intervention (No Intervention): The control group will not participate in any intervention for the duration of the study. In addition, the participants will be instructed to follow their usual daily schedule for 6 months. Changes in health, medication, or habits will be discussed by the investigators' team and reassess the continuation or the termination of the investigated participant.
- Lifestyle Medicine Strategies Groupo (Experimental): The LSM (LifeStyle Medicine) group, will receive a 6-month lifestyle change intervention targeting the correction of diet, improving physical activity and exercise levels, reducing stress levels, and improving sleep hygiene by LSM registered professionals.
  Interventions: Behavioral: Lifestyle Medicine Strategies

INTERVENTIONS:
Behavioral: Lifestyle Medicine Strategies — LM addresses health risk factors in primary, secondary, and tertiary prevention of developing disease rather than limiting resources and medical expenditures on acute care and reacting to illness, injury, and disease.
  The intervention will target the four pillars of the LM approach including physical activity, diet, stress, and sleep. Certified in LM strategies professionals will consult participants from the LM group in a biweekly base in order to improve their lifestyle habits.
  Arms: Lifestyle Medicine Strategies Groupo

SUMMARY:
Sleep has a number of health benefits, including memory and learning, vitality and energy as well as high quality of life levels. Lack of sleep impairs judgment, impacts longevity and safety, and increases the risk of a number of diseases including obesity, hypertension, heart disease, diabetes, mood disorders, and impaired immune function. In addition lack of sleep or disturbance of normal sleep cycle could have a major impact on people's lives and working performance such as driving. Daily sleepiness is a problem concerning professions with a non-fixed schedule. Specifically, professional long-haul drivers confront sleepiness problems and in combination with fatigue, they are prone to driving accidents and other incidents. Sleep quality and quantity are closed related to fatigue which is one of the most common reasons for driving and working accidents. In recent years, car accidents involving professional drives have increased significantly. The main reasons for those accidents were fatigue and sleepiness due to long hours of driving or difficult working conditions according to the recent European report (Driver Fatigue in European Road Transport - etf-europe.org).

Lifestyle Medicine addresses health risk factors in primary, secondary, and tertiary prevention of developing disease rather than on acute care and reacting to illness, injury, and disease. Lifestyle Medicine strategies targeting modifiable risk factors, such as diet, sleep, stress, and physical activity. By applying those regimes the investigators could improve physical and mental health levels that can affect the quality of sleep, reducing daily sleepiness and fatigue, in professional drivers operating coaches and trucks. Any intervention that could improve alertness and reduce fatigue and sleepiness in those people, will automatically improve safety, reduce driving accidents and save lives and resources.

DETAILED DESCRIPTION:
Methodology Participants: Professional divers with valid 5th category driving license will be the target group of this RCT. All participants will sign an informed consent form in order to participate in the study. Participants will undergo a complete health history and will have the approval of their attending physician. The study has been approved by the local IRB Internal Ethics Committee.

Study Design: This is a randomized clinical trial involving healthy human volunteers. Participants will be assessed before and after a 6-month lifestyle intervention. The current project consists of 9 interconnected Steps:

Step 1: Participants will sign the consent form and complete the PARQ health questionnaire for assessing the readiness to exercise participation followed by the Epworth Sleepiness Scale (SSC) for assessing daily sleepiness.

Step 2: Participants that fulfill the inclusion criteria will be scheduled for a full night Polysomnography test at the sleep unit of the Center of Research and Evaluation of Human Performance (CREHP) laboratory.

Step 3: After completing the polysomnography test, participants will complete a 2h OGTT test for assessing insulin resistance and glucose tolerance. During those two hours, the participants will complete a series of questionnaires assessing aspects related to demographics, quality of life, health, and sleep quality.

Step 4: After the completion of Step 3, participants will go through a body composition analysis using the DEXA method followed by a bioimpedance analysis for assessing total body water levels.

Step 5: After the completion of Step 4, participants will participate in a battery of tests assessing fitness levels and functional capacity. Physical activity levels will be recorded using a mobile application for the duration of a week.

Step 6: After the completion of Step 5, participants will be scheduled after 2 days for a lab Multiple Sleep Latency Test (MSLT) for the assessment of their levels of daily sleepiness.

Step 7: After the completion of Step 6, participants will follow a series of interviews with certified experts. More specifically,

* a registered dietitian will assess nutritional habits and prescribe a corrective diet in order to improve the participants' nutritional profile.
* a registered psychologist will assess mental health and stress levels and suggest corrective approaches for improving participants' stress levels and mental capacity.
* a registered exercise physiologist will assess fitness levels and prescribe an appropriate exercise training program for improving cardiovascular fitness and functional capacity.
* a registered sleep coach will assess sleep quality and hygiene and suggest ways for improving sleep quality and restfulness.

Step 8: After completion of Step 7 participants will be given a 24h Blood Pressure (BP) Holter for assessing the circadian variation of BP and a Heart Rate Variability (HRV) monitor for assessing HRV during a normal working day (including driving).

Step 9: After the completion of all steps, participants will be randomly assigned to one of the two groups based on demographic and sleep parameters: the control group (CON) and the experimental group (EXP).

Intervention: The intervention of the current project includes 6 months of lifestyle modification counseling based on the guidelines and principles of the European Lifestyle Medicine Organization (eulm.org). More specifically, counseling will target areas such as nutrition, exercise, stress, and sleep. A certified specialist will interview and assess all participants and prescribe the appropriate corrective regimes for improving participants' lifestyles and reducing cardiovascular risk factors. More particularly, for nutritional counseling a customized diet will be provided and change every two weeks, for exercise counseling, a customized supervised exercised training will be provided and change every two weeks, for psychological counseling, a customized psychological approach will be provided and reassessed every two weeks and for sleep counseling, a customized sleep hygiene program will be provided and reevaluated every month.

Randomization: Randomization will take place using a randomization computer software. Randomization will consider parameters such as gender, age, BMI, and sleepiness score.

Measurements:

Demographic Characteristics: Demographic characteristics include age, gender, race/ethnicity, education, socioeconomic status, health, disability status, and work-related information.

Questionnaires: Various validated questionnaires will be used for the assessment of aspects related to the quality of life and health using the interview method.

General Health: The PARQ questionnaire will be used for the assessment of the level of readiness to participate in an exercise training program. The General Health Questionnaire 30 (GHQ30) will be used for the assessment of the general health status of the participants. Charlson Comorbidity index will be used for the calculation of the comorbidity index.

Sleepiness and Quality of Sleep: The Epworth Sleepiness Scale (ESS) will be used for the assessment of the level of sleepiness. The Pittsburgh Sleep Quality Index (PSQI) will be used for the assessment of sleep quality and sleep abnormalities. Furthermore, the Karolinska Sleepiness Scale (KSS) will be used for the assessment of alertness and vitality. Finally, the Daily Sleep Diary will be used for the assessment of the level of sleep quality of the participants.

Fatigue levels: The Fatigue Severity Scale (FSS) will be used for the assessment of the level of general fatigue.

The quality of life: The SF36QoL questionnaire (SF-36) will be used for the assessment of the levels of quality of life.

Depressive symptoms: The Beck Depression Inventory (BDI) questionnaire will be used for the assessment of depressive symptoms and signs.

Stress: The Perceived Stress Scale (PSS) and the Work Stress Questionnaire (WSQ) will be used for the assessment of stress levels.

Physical Activity: The International Physical Activity Questionnaire (IPAQ) will be used for the assessment of physical activity levels.

Driving Skills and Habits: The Driving Habits Questionnaire (DHQ) will be used for the assessment of driving habits.

Nutrition: The General Nutrition Knowledge Questionnaire (GNKQ) will be used for the assessment of nutritional knowledge and habits.

Biochemical Analysis: Blood samples will be collected after overnight fasting for measurement of lipids, hormones, and general hematology analysis. Glucose disposal and indices of insulin resistance will be assessed by an Oral Glucose Tolerance Test (Blood samples will be collected 0, 30, 60, 90, and 120 minutes following ingestion of 75gr of glucose). The insulin resistance index will be calculated by the OGIS and HOMA-IR equations.

Body Composition: Body composition will be assessed using anthropometric measurements including BMI, WHR as well as DEXA scans for the assessment of total and regional fat and lean body mass (Lunar model DPX Madison, WI). Intracellular and extracellular as well as total body water levels will be measured by bioimpedance using a portable BIA system, (Tanita BC 543).

Blood Pressure: The circadian blood pressure variation will be assessed using a 24h BP Holter (GIMA 24HABPM).

Heart Rate Variability: Heart Rate Variability will be assessed using a portable ECG designed to measure all HRV indices (OMRON HCG-801).

Sleep Quality Assessment: Quality and quantity of sleep will be assessed by an overnight Polysomnographic study (PSG). Levels of daily sleepiness will be assessed using the Multiple Sleep Latency Test (MSLT). MSLT is a full-day test that consists of five scheduled naps separated by two-hour breaks.

Fitness Assessment Physical Activity: A mobile phone-based steps tracking application will be used for the assessment of the weekly physical activity levels.

Aerobic Capacity: The six-minute walk test (6MWT) will be used for the assessment of Aerobic capacity and Endurance.

Strength: 1RM will be used for the assessment for the evaluation of maximum muscle strength. Also, the sit to stand-60sec (STS60) test will be used for the assessment for testing leg strength and endurance. Finally, a 5x sit-to-stand test (STS5) will be used for the assessment of functional lower extremity strength, transitional movements, balance, and fall risk.

Flexibility: The Sit and Reach test (S&R) will be used for the assessment of flexibility of the lower back and hamstring muscles.

Handgrip: The handgrip test will be used for the assessment of the maximum isometric strength of the hand and for arm muscles (Marsden MG-4800 Hand Dynamometer).

Statistics SPSS statistical software (SPSS 21, Illinois USA) will be used for statistical analysis.

The pre and post within Control (Con) and Exercise (Ex) groups will be examined by using paired t-test. Correlations between (Con) group and (Ex) group parameters will be examined by using Spearman correlation. Also, will be examined Δ change values by using an unpaired t-test.

Power Analysis:

Power analysis was performed using the open-source software G*Power (3.1.9.2) and was used to calculate the minimum number of participants required to achieve reasonable power (>85%). A priori compute required sample size analysis revealed that in one of the main parameters related to the aims of the study (ESS score), the study needs a total sample size of 42 participants (for both groups) in order to have enough power to detect statistically significant differences between the pre and post-intervention comparisons (within groups ESS: Effect size dz=0.4783, total sample size=42, t=2.019, Power (1-β err prob)=0.88289). Given an estimation of a reasonable dropout rate of 20%, it is estimated that a number of 25 participants per group is needed in order to have significant power to achieve meaningful results.

ELIGIBILITY:
Inclusion Criteria:

* both sexes,
* age between 25 and 60 yrs old
* valid 5th category driving license for large trucks and coaches
* minimum of 3 years of continuous and verifiable documented work experience as a professional driver in the past 5 years
* diagnosed with moderate daily sleepiness as this is documented by a value >9 in Epworth Sleepiness Scale (SSC)

Exclusion Criteria:

* drivers with a driving license that expires within a year of the recruitment date,
* disabilities that prevent them from walking independently or exercising,
* verified mental illnesses,
* alcoholism or drug abuses,
* or conditions that could affect the outcome of the study

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in Daily Sleepiness | Assessed at 0-month (pre) and at 6-month (post)
  The levels of daily sleepiness will be assessed by a Multiple Sleep Latency Test (MSLT). This is the gold standard approach for assessing daily sleepiness.
Changes in Levels fo Fatigue | Assessed at 0-month (pre) and at 6-month (post)
  The levels of fatigue will be assessed by the FSS test
Changes in Quality of Sleep | Assessed at 0-month (pre) and at 6-month (post)
  Quality of sleep will be assessed by a full night polysomnography study

SECONDARY OUTCOMES:
Changes in Body composition | Assessed at 0-month (pre) and at 6-month (post)
  The changes in body composition will be measured by the DEXA method
Changes in Exercise Capacity | Assessed at 0-month (pre) and at 6-month (post)
  Exercise capacity will be assessed by 6 min walk test
Changes in Stress levels Work Stress Questionnaire | Assessed at 0-month (pre) and at 6-month (post)
  Stress levels will be assessed by validated questionnaires.
Changes in Quality of Life levels | Assessed at 0-month (pre) and at 6-month (post)
  Quality of life will be assessed by SF36 QoL questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgos K Sakkas, PhD, Principal Investigator — University of Thessaly; Efthmios Dardiotis, MD, PhD, Study Chair — University of Thessaly
Locations (1):
- Lifestlye Medicine Laboratory, TEFAA, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No